CLINICAL TRIAL: NCT01984333
Title: Developing Online Response Inhibition Training for Individuals With Trichotillomania
Brief Title: Online Response Inhibition Training for Trichotillomania
Acronym: OTTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Han Joo Lee, Assistant Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UWMRF-133
Record Dates: First submitted 2013-11-01; First posted 2013-11-14 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Trichotillomania
Keywords: trichotillomania; response inhibition; cognitive retraining
MeSH Terms: conditions — Trichotillomania

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online cognitive training (Experimental): Online cognitive training will provides eight sessions of a computerized training game. Each session will last about 30-40 minutes, and participants will undergo 2 sessions each week over a 4-week period.
  Interventions: Behavioral: Online cognitive training
- Waitlist control (No Intervention): This is a 1-month waitlist control to be compared with the active online cognitive training intervention. This is a no intervention control group.

INTERVENTIONS:
Behavioral: Online cognitive training — Online cognitive training is a web-based video game that offers systematic training of response inhibition capabilities. Participants will be guided to make progress in an individually-tailored fashion to master increasingly difficult game levels.
  Arms: Online cognitive training

SUMMARY:
Trichotillomania (TTM) remains one of the most poorly-understood and inadequately-treated conditions. Research has shown poor response inhibition (RI; the ability to inhibit inappropriate but potent response) as an important cognitive feature of TTM. Investigators have developed a computerized training program that aims to improve RI. Fifty children with TTM will be randomly assigned to (a) online 8-session RI training (n=25), or (b) 1-month waitlist condition (n = 25), and will be assessed at baseline, post-treatment, and 1-month follow-up. Investigators hypothesize that the online RIT will show greater improvement in TTM symptoms and RI capabilities at post-treatment and 1-month follow-up assessments, compared to the waitlist condition. This study will help develop an effective cognitive intervention program for TTM.

DETAILED DESCRIPTION:
Although trichotillomania (TTM), an impulse control disorder characterized by compulsive hair pulling, typically results in serious consequences including impaired individual functioning, medical problems (e.g., skin infections), and elevated comorbidity with other psychiatric disorders, it remains one of the most poorly-understood and inadequately-treated psychiatric conditions. There is an urgent need for effective and accessible clinical interventions for TTM, especially for young individuals who suffer from a marked lack of adequate treatment resources despite the early onset of the condition. One promising therapeutic approach is to improve cognitive problems believed to contribute to TTM, using a computerized cognitive retraining method. Research has indicated impaired response inhibition (RI; the ability to inhibit inappropriate but potent response) as an important cognitive feature underlying TTM. Therefore, RI is considered to be an important target of cognitive retraining. Investigators have developed a computerized training program that aims to improve RI capabilities in the format of an online video game. Fifty children with TTM will be randomly assigned to (a) online 8-session RIT (n=25), or (b) 1-month waitlist condition (n = 25), and will be assessed at baseline, post-treatment, and 1-month follow-up. The waitlisted participants will also be invited to undergo the training program after the 1-month follow-up assessment is completed. Investigators hypothesize that the online RIT will show greater improvement in TTM symptoms and RI capabilities at post-treatment and 1-month follow-up assessments, compared to the waitlist condition. This study is expected to generate important data that will guide the development of an accessible, cost-efficient, and effective cognitive intervention for individuals suffering from TTM.

ELIGIBILITY:
Inclusion Criteria:

* age between 8 and 17
* a diagnosis of trichotillomania
* a computer with high speed internet

Exclusion Criteria:

* current substance use problems
* current or past psychotic disorder, bipolar disorder, or schizophrenia
* current behavioral treatments for trichotillomania
* significant suicidality
* severe conditions known for poor response inhibition(ADHD, OCD, and tic disorders)
* recent or planned change in medication
* low intellectual functioning (below 80)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2013-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change on the NIMH Trichotillomania Severity and Impairment Scales | Baseline, 4 weeks, and 1-month Follow-up
  These are clinician-rated measures for assessing the severity of trichotillomania and the impairment caused by hair pulling. This measure will be administered at baseline, at 4 weeks, and at 1-month follow-up.

SECONDARY OUTCOMES:
Change on the Clinical Global Impression Scale | Baseline, 4 weeks, and 1-month Follow-up
  This is a widely used brief assessment tool for evaluating illness severity, global improvement or change, and therapeutic response. This measure will be administered at baseline, at 4 weeks, and at 1-month follow-up.

OTHER OUTCOMES:
Change on the Trichotillomania Scale for Children | Baseline, 4 weeks, and 1-month Follow-up
  This is a widely used self-report measure of hair pulling symptoms. Both the participant and parent will fill out this questionnaire at baseline, at 4 weeks, and at 1-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Hanjoo Lee, Ph.D., Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- UWM Anxiety Disorders Laboratory, Milwaukee, Wisconsin, United States